CLINICAL TRIAL: NCT02901262
Title: Utility of Continuous Electroencephalogram and Derived Variables in NeuroIntensive Care
Brief Title: Continuous Quantified EEG in NeuroIntensive Care
Acronym: CrazyEEG
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera San Gerardo di Monza (Other)
Collaborators: Papa Giovanni XXIII Hospital (Other)
Responsible Party: Principal Investigator, Prof. Giuseppe Citerio, NeuroIntensive Care Director, Azienda Ospedaliera San Gerardo di Monza
Other Study IDs: EEG2016
Record Dates: First submitted 2016-08-19; First posted 2016-09-15 (Estimated); Results first posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2023-09

CONDITIONS: Coma; Traumatic Brain Injury; Subarachnoid Hemorrhage; Ischemic Stroke
Keywords: continuous EEG
MeSH Terms: conditions — Coma; Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- qEEG patients: All the patients with continuous EEG (>24 hours) in the two study units

SUMMARY:
To evaluate the ability of NICU (NeuroIntensive Care Unit) staff to interpret, before and after a training period, symmetry, sedation level, seizures activities and artefact on continuous cEEG/qEEG (continuous electroencephalography/quantitative electroencephalography) tracings.

DETAILED DESCRIPTION:
Using a web based tool, the clinicians of the two study centers will review 24 hours of recording (raw EEG data + derived qEEG variables).

The intensivists will evaluate:

* simmetry,
* sedation level,
* seizures activities and
* artefact on continuous cEEG/qEEG tracings. The same tracings will be blindly reviewed by a certified neurophysiologist (using the app). The neurophysiologist evaluation will be considered as "reference".

The results of the evaluation will be compared (intensivists vs. neurophysiologist) in order to understand if the intensivists are able to adequately identify the pathological findings.

The study period will be:

* before a formal training
* after a formal training by neurophysiologist in order to understand if the training is able to improve the intensivists performance.

ELIGIBILITY:
Inclusion Criteria:

Intensivists wil evaluate daily qEEG recordings of:

* Patients in coma after a traumatic/vascular event
* Admitted to neurointensive care and
* Recorded with continuous EEG for clinical reasons

Exclusion Criteria:

* No EEG recording > 24 hours

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Intensivists will evaluate tracing from patients in coma after a traumatic/vascular event admitted to neurointensive care and recorded with continuous EEG for clinical reasons
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Citerio, MD, Principal Investigator — Università Milano Bicocca
Locations (2):
- Italy (2):
  - Azienda Ospedaliera Papa Giovanni Xxiii, Bergamo
  - Azienda Ospedaliera San Gerardo, Monza

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After the evaluation of qEEG (quantitative electroencephalography) from 30 patients, other intensivists and neurophysiologists were engaged to use the customized web-based online application that was downloaded on computers and cell phones to evaluate qEEG.
Units Other Than Participants: qEEG evaluations
Groups:
- Study Cohort: From February to August 2016 periods of >12 h of cEEG (continuous electroencephalography) were independently evaluated by intensivists and by neurophysiologists using a customized web-based online application that was downloaded on computers and cell phones. A total of 86 paired evaluations were performed in 30 patients, and 1740 h of qEEG (quantitative electroencephalography) was subsequently evaluated.
Period: Overall Study
Arm/Group | Study Cohort
Started | 30; 86 qEEG evaluations
Completed | 30; 86 qEEG evaluations
Not Completed | 0; 0 qEEG evaluations

BASELINE CHARACTERISTICS:
Arm/Group | qEEG Patients
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 30

OUTCOME MEASURES:

1. Primary Outcome: Number of Correct qEEG Evaluations
Description: Percentage of correct evaluation of qEEG tracings by intensivists vs. neurophysiologist.
  The result will be expressed as percentage of correct evaluations for each domain.
Time Frame: 2 months
Population: Neuro-intensivists, after the in-house training
Measure: Number; unit: percentage of correct evaluation
Units Other Than Participants: qEEG evaluations
Groups:
- Study Cohort: From February to August 2016 periods of >12 h of cEEG were independently evaluated by intensivists and by neurophysiologists using a customized web-based online application that was downloaded on computers and cell phones. A total of 86 paired evaluations were performed in 30 patients, and 1740 h of qEEG was subsequently evaluated.
Arm/Group | Study Cohort
Number analyzed (Participants) | 30
Number analyzed (qEEG evaluations) | 86
percentage of correct evaluation
  Simmetry | 70
  Sedation level | 78
  Seizures activities | 69
  artefact on continuous cEEG/qEEG tracings | 82

2. Secondary Outcome: Kappa Coefficient of Agreement Between Intensivists and Neurophysiologists After Training
Description: Comparison of the correct answers of the intensivist before and after a period of training.
  Results will be expressed as coefficient of agreement between neurophysiologists and intensivists in interpretation of the tracings of continuous electroencephalography using Cohen's kappa coefficient, after training
Time Frame: 12 months
Population: Agreement between neurophysiologists and intensivists in interpretation of the tracings after training
Measure: Mean (95% Confidence Interval); unit: Kappa Coefficient
Units Other Than Participants: qEEG evaluations
Arm/Group | Study Cohort
Number analyzed (Participants) | 30
Number analyzed (qEEG evaluations) | 86
Kappa Coefficient
  Seizures | 0.5 [0.3 to 0.7]
  Simmetry | 0.65 [0.5 to 0.8]
  Artefacts | 0.6 [0.4 to 0.8]
  Sedation | 0.75 [0.55 to 0.9]

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed
Groups:
- qEEG Patients: All the patients with continuous EEG (>24 hours) in teh two study units
Arm/Group | qEEG Patients
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes